CLINICAL TRIAL: NCT02459015
Title: A Controlled, Randomized, Comparison, Blind Evaluation of Repair of Digital Nerve Lesions in Man Using an Implanted Reaxon® Nerve Guide
Brief Title: Performance Study of an Artificial Nerve Guide (Reaxon® Nerve Guide) to Treat Digital Nerve Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to slow patient recruitment and insufficient patient compliance.
Sponsor: Medovent GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NG-001
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Reaxon® Nerve Guide (Experimental): Implantation of Reaxon® Nerve Guide: If the subject is randomized to the Reaxon® Nerve Guide group, the surgeon will implant a Reaxon® Nerve Guide of ≤ 30 mm to bridge a nerve defect of ≤ 26 mm according to the method described in the instructions for use.
  Interventions: Device: Implantation
- Autologous Nerve Graft (Active Comparator): Implantation of an autologous nerve graft: If the subject is randomized to the conventional treatment, the surgeon will repair the nerve by interposing an autologous nerve graft of ≤ 26 mm between the nerve ends.
  Interventions: Device: Implantation

INTERVENTIONS:
Device: Implantation — A peripheral nerve defect up to 26 mm in the finger will be repaired by implantation of either a Reaxon® Nerve Guide or an autologous nerve graft (depending on the randomization group) on day 0.

SUMMARY:
The purpose of this clinical investigation is to confirm the medium- and long-term safety and performance of the chitosan-based nerve guide (Reaxon® Nerve Guide) in comparison to an autologous nerve graft to bridge nerve defects in the finger.

DETAILED DESCRIPTION:
The clinical investigation NG-001 is a multicenter, parallel, controlled, randomized, blind evaluation of the repair of digital nerve lesions.

Medovent will perform this clinical investigation as a post-market clinical follow-up (PMCF) study in accordance with the MEDDEV 2.12/2 rev2 guidelines to confirm the medium- and long-term safety and performance of its chitosan-based nerve guide (Reaxon® Nerve Guide). The results of this investigation will be used by Medovent to update the clinical evaluation throughout the life-cycle of Reaxon® Nerve Guide and to ensure its long term safety and performance in the market. Additionally, Medovent will include the application of Reaxon® Nerve Guide in digital nerves to confirm the safety of applying Reaxon® Nerve Guide over joints.

The study will be performed in specialized German centers. A total number of 76 subjects with traumatic digital nerve injuries in whom surgical repair may not allow end-to-end direct suture of the nerve ends, and in whom the nerve tissue gap would indicate the use of an autograft of equal or less than 26 mm, are eligible for inclusion.

The primary objective of the clinical investigation is to demonstrate that the static 2-point discrimination (2-PD) 12 months after surgery will be not inferior in the Reaxon® Nerve Guide test group compared to the control group receiving an autologous nerve graft.

The secondary objective is to document the long-term effects (up to 18 months after surgery) in nerve repair. The non-inferiority test is to demonstrate that it can be excluded that the treatment difference is larger than 20% in favor for the control group.

ELIGIBILITY:
Inclusion Criteria:

1. males and females between 18 and 65 years of age able to give his/her consent
2. a complete traumatic nerve injury of the common or proper digital nerve in the hand
3. a nerve defect of less or equal than 26 mm after release and approximation of the nerve ends and measured when the wrist is in neutral position
4. an injury that could conventionally be treated with implantation of a short nerve graft
5. nerve treatment initiated until 3 months after nerve injury
6. signed informed consent

Exclusion Criteria:

1. known allergy to chitosan and/or polyvinylpyrrolidone (PVP)
2. known impairment / previous diseases of the neural axis or previous lesions of the affected hand (of the digital nerve), which led to permanent sensory or motor restrictions of the hand/finger
3. complete amputation injury
4. known pregnant or breast-feeding females
5. disorders known leading to impaired wound healing (e.g. diabetes mellitus)
6. skin diseases in the wound area
7. impaired blood coagulation or bleeding disorders (e.g. because of regular intake of cumarin such as Marcumar)
8. pathologic blood flow disorders (e.g. Morbus Raynaud)
9. participated in another clinical investigation using an investigational new drug or device within 30 days prior to enrolment into this investigation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-06; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Static 2-point discrimination (2-PD) | Primary outcome analysis will be performed from the clinical evaluations at 12 months post-surgery
  The perception of either one or two points of touch is assessed using a small tool with prongs at fixed spacing's from 2 to 15 mm. One or two points will be applied randomly in a longitudinal direction on the distal phalanx of all fingers.
  Grades/scores:
  0 = > 15 mm (poor)
  1. = 11-15 mm (fair)
  2. = 6-10 mm (good)
  3. = < 6 mm (excellent)
  Scores of 2 or 3 will be evaluated as (meaningful) response. At a score of 0 it will further be determined if the subject has protective sensibility or is anesthetic. A disposable cannula can be used.
  Single point is noticeable = protective sensibility No point is noticeable = anesthetic

SECONDARY OUTCOMES:
Static 2-point discrimination (2-PD) | Baseline visit (latest 7 days post-surgery) + Follow-up examinations 3, 6, 12 and 18 months post-surgery
  see description above
Moving 2-PD | Baseline visit (latest 7 days post-surgery) + Follow-up examinations 3, 6, 12 and 18 months post-surgery
  A moving stimulus of either one or two points is assessed using a small tool with prongs at fixed spacing's from 2 to 15 mm. One or two points will be moved randomly in a longitudinal direction from proximal to distal of all fingers.
  Grades/scores: see Static 2-PD
Semmes-Weinstein Monofilament | Follow-up examinations 3, 6, 12 and 18 months post-surgery
  The 5 kit monofilaments will be used. A monofilament is pressed against the skin at specific locations (see protocol) starting with the thinnest filament (i.e. 2.83) and then, depending on the response, thicker filaments are applied until the subject feels the pressure.
  Grades/scores:
  0 = not testable
  1. = filament 6.65, perception of deep pressure
  2. = filament 4.56, no protective sensation
  3. = filament 4.31, diminished protective sensation
  4. = filament 3.61, diminished perception of light touch
  5. = filament 2.83, normal perception of light touch
Subject's estimation of cold intolerance and hyperesthesia | Follow-up examinations 3, 6, 12 and 18 months post-surgery
  The examiner will stroke the dysfuntional area and question the subject about cold intolerance and hypersensitivity.
  Grades/scores:
  0 = Hinders function
  1. = Disturbing
  2. = Moderate
  3. = None/minor
Hoffmann-Tinel-Test | Follow-up examinations 3, 6, 12 and 18 months post-surgery
  The test is performed by lightly tapping over the nerve to elicit a sensation of tingling in the distribution of the nerve. The distance of the sensation from the distal end of the implant will be determined.
post-operative complications | Baseline visit (latest 7 days post-surgery) + Follow-up examinations 3, 6, 12 and 18 months post-surgery
  There will be evaluations of common post-operative complications associated with peripheral nerve repair surgery, i.e. painful neuroma formation, assessed by pain on percussion, allodynia, and dysaesthesia (pain and/or numbness).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Siemers, PD Dr. med., Principal Investigator — BG-Kliniken Bergmannstrost
Locations (4):
- Germany (4):
  - BG-Kliniken Bergmannstrost, Halle, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Unfallkrankenhaus Berlin, Berlin
  - BG Kliniken Hamburg gGmbH, Hamburg